CLINICAL TRIAL: NCT02522312
Title: A Retrospective Analysis of Restasis® Benefits in Dry Eye Contact Lens Patients
Status: Completed | Type: Observational
Sponsor: Hazleton Eye Specialists (Other)
Responsible Party: Principal Investigator, Dr. Thomas P. Kislan, Doctor at and Owner of Hazleton Eye Specialists, Hazleton Eye Specialists
Other Study IDs: IIT-00864
Record Dates: First submitted 2015-07-29; First posted 2015-08-13 (Estimated); Last update posted 2016-03-03 (Estimated); Status verified 2016-03

CONDITIONS: Dry Eye Syndrome
Keywords: Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: No Intervention — No drug is administered in this study

SUMMARY:
A retrospective analysis of Restasis® benefits in dry eye contact lens patients.

DETAILED DESCRIPTION:
Charts of contact lens wearers with diagnosed dry eye who are being treated with Restasis will be evaluated to determine success in treatment by retrospectively looking at various outcome measures including but not limited to schirmer, staining and osmolarity levels

ELIGIBILITY:
Inclusion Criteria:

* Male or Female, > or = 18 years of age
* Subject was previously diagnosed (prior to Baseline Visit) with mild to severe dry eye disease (ITF level 1, 2 or 3) which required continuous medical therapy with Restasis® for a minimum duration of 6 months post-Baseline (Visit 1); or Subject was newly diagnosed (at Baseline Visit) with mild to severe dry eye disease (ITF level 1, 2 or 3) which required continuous medical therapy with Restasis® for a minimum duration of 6 months post-Baseline (Visit 1);
* Subject was prescribed Restasis® therapy at Baseline Visit (Visit 1) and commenced dosing immediately after Baseline Visit (Visit 1)
* Baseline Visit occured between 01 July 2012 and 01 January 2014;
* Subject had corneal staining and at least one dry eye sign (i.e., Schirmer's Test score <10 mm, decreased tear lake, TBUT <10 seconds, conjunctival staining, tear osmolarity >310 mOsmol/L
* Subject had charted tolerability and efficacy data reflecting at least one follow-up visit following Restasis® treatment initiation; and
* Subject wore contact lens(es) concurrently while receiving Restasis® treatment for a minimum duration of 6 months post-Baseline (Visit 1)

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary Care Clinic
Sampling Method: Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2015-09; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Improvement of Schirmer's Test score | 6 months
Increased contact lens wear time | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Thomas P Kislan, Dr., Principal Investigator — Owner
Locations (1):
- Hazleton Eye Specialists, Hazleton, Pennsylvania, United States